CLINICAL TRIAL: NCT05191095
Title: The Accuracy of Human Endoscopic Detection of Submucosal Invasive Cancer in Colorectal Polyps - Analysis of 739 Individual Assessments of Large Non-pedunculated Colorectal Polyps Using a Novel Clinical Decision Support Tool
Brief Title: The Accuracy of Human Endoscopic Detection of Submucosal Invasive Cancer in Colorectal Polyps
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-09381 + E01
Record Dates: First submitted 2021-11-23; First posted 2022-01-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Polyp

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Colorectal cancer (CRC) is a leading cause of death in the Western world. It can be effectively prevented by removal of pre-malignant polyps (polypectomy) during colonoscopy. Large (≥20mm) non-pedunculated colorectal polyps (LNPCPs) represent 2-3% of colorectal polyps, and require special attention prior to treatment. If submucosal invasion (SMI) is suspected careful decision making is required to exclude features which unacceptably increase the risk of lymph node metastases and render local treatment (endoscopic) non-curative. Such patients require a multi-disciplinary approach and consideration of surgery +/- systemic therapy.

Recently the endoscopic imaging characteristics which precisely determine the risk of SMI within colon polyps have been elucidated. This suggests endoscopic imaging may be the ideal investigation to stratify the presence and extent of SMI within LNPCP, particularly as it can be applied in real-time at the time of planned endoscopic treatment.

Unfortunately, current classification systems are complex, require extensive training and technology not available in the majority of non-tertiary hospitals. They are therefore underused leading to incorrect decision making and negative patient outcome (e.g piecemeal resection without the chance of endoscopic cure or unnecessary further procedures in referral centres with resultant surgery anyway or surgery for benign disease)

A simple clinical support tool was created, based on well-established parameters (i.e., presence of a demarcated area within a polyp, size of the polyp, Paris classification, location within the colon and granularity) to identify OVERT (visible on the surface) and COVERT (hidden) submucosal invasion (SMI) within LNPCPs. Crucially this tool only uses what is reproducible in the majority of endoscopy units in the Western world (i.e. standard magnification, no extra chromic dyes etc). predict SMI within LNPCPs and we translated it into a single web-based clinical support tool that can be used by every endoscopist (expert and non-expert).

To evaluate the tool, a survey will be send to participants. The survey consist of a 10-minute educational video where the use of the tool will be explained. Then 20 standardised videos of LNPCPs will be shown. Participants are first asked about their first impression regarding the presence of SMI. Then they are redirected to the web-based tool. After filling the required data from a standardised video (45 seconds to minute, no focus on one particular area of the polyp) the score generated by our tool is copied to the participants computer clipboard and then pasted in the survey so that we could analyse it.

ELIGIBILITY:
Inclusion Criteria:

* Gastrointestinal endoscopic experience (trainees, student, gastroenterologist consult, surgeon)

Exclusion Criteria:

* No connection with endoscopy in gastroenterology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We study the accuracy of human detection of submucosal invasive cancer within colorectal polyps amongst endoscopist of varying experience
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
The accuracy of endoscopic assessment as to the risk of SMI within LNPCPs from a standardised endoscopic video, using a novel, freely accessible, web-based simple clinical decision support tool as versus expert opinion. | 30 minutes
  Can participants, using the tool, identify SMI within LNPCPs?

SECONDARY OUTCOMES:
The inter-observer agreement of a novel simple clinical decision support tool to determine the risk of SMI within LNPCPs from a standardised endoscopic video as versus expert opinion. | 30 minutes
  Are participants able to derive characteristic information from polyps (size, Paris classification, granularity, pit/vascular pattern) using a standardised video of LNPCPs

CONTACTS AND LOCATIONS:
Overall Officials: David Tate, Principal Investigator — UZ Gent
Locations (1):
- UZ Gent, Ghent, Belgium